CLINICAL TRIAL: NCT03976635
Title: Evaluation of Pain, Discomfort and Acceptance During the Orthodontic Treatment of Class III Malocclusion Using Bone-anchored Intermaxillary Traction Versus the Removable Mandibular Retractor: A Randomized Controlled Trial
Brief Title: Evaluation of Pain, Discomfort and Acceptance During the Orthodontic Treatment of Class III Malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Collaborators: Hama University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-01-2019
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Class III Malocclusion; Cross Bite; Orthodontic Appliance Complication
Keywords: Removable Mandibular Retractor; Bone-anchored Intermaxillary Traction
MeSH Terms: conditions — Malocclusion, Angle Class III; Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Removable Mandibular Retractor (Active Comparator): Patients in this group will be treated by the Removable Mandibular Retractor (RMR) in order to get rid of the anterior cross bite. This appliance is removable.
  Interventions: Device: Removable Mandibular Retractor
- Bone-anchored intermaxillary Traction (Experimental): Patients will be treated using bone-anchored intermaxillary traction. Class III elastics will be extended from the Adam's clasps placed in the upper removable appliance towards the heads of mini-implants placed between the permanent canine and lateral incisors on either side of the lower dental arch.
  Interventions: Device: Bone-anchored intermaxillary traction

INTERVENTIONS:
Device: Removable Mandibular Retractor — The appliance will be used 18 hours per day. It can only be removed for eating meals.
  Other Names: RMR; Inferiorly extended labial bow; Reverse Hawley bow
  Arms: Removable Mandibular Retractor
Device: Bone-anchored intermaxillary traction — The patients will be instructed to wear the upper removable appliance for 18 hours per day. The elastics should be extended from the upper appliance towards the lower mini-screws.
  Other Names: BAIMT
  Arms: Bone-anchored intermaxillary Traction

SUMMARY:
The aim of this study is to evaluate the levels of pain, discomfort and acceptance between two treatment modalities of Class III correction of growing patients in the late mixed dentition period.

DETAILED DESCRIPTION:
The acceptance of orthodontic appliance is measured by the amount of discomfort occurring during orthodontic treatment. Different feelings can be encountered during the course of orthodontic treatment such as pressure, tension and pain. Pain is defined as an unpleasant feeling and a bad subjective experience combined with internal or external reason and it is considered as the most annoying factor during orthodontic treatment with fixed appliance. In a study by Oliver and Knappman, patients stated that the worse thing related to the orthodontic treatment was pain and 70% of the subjects suffered from pain during orthodontic treatment regardless the appliance' type. The fear from the pain is considered as the most important factor that not encourage patient to ask orthodontic treatment.Many studies demonstrated that there were no differences in the amount of the pain resulted from the orthodontic treatment between males and females [2, 5]. In a study of the reasons which make patient stopped the orthodontic treatment, Haynes found that the pain was the first reason, whereas the second one was the effect of the orthodontic appliance on the patient's daily social life.

When reviewing the medical literature, few studies have been found to identify the patient acceptance degree to the orthodontic appliance used for treating Class III cases in general and Class III functional appliances in particular.Removable appliances were evaluated by a series of publications by Sergl et al in Germany.Additionally, when rigorous study designs are considered utilizing randomized controlled trials (RCTs), there are only few RCTs in the dental literature that evaluated patients' responses towards orthodontic treatment. Idris et al., evaluated Class II growing patients undergoing functional orthopedic corrections, whereas Khattab et al., compared labial brackets versus lingual brackets in terms of speech and functional impairments. Recently, Saleh et al., evaluated the levels of acceptance towards the removable mandibular retractor (RMR) when treating young children with Class III malocclusion in the late primary dentition and early mixed dentition (i.e. between 5 and 9 years) and found high levels of acceptance recommending the need for further analysis of patients' responses to this appliance in older age groups.

Bone-anchored intermaxillary elastics have been proposed as a method of correcting Class III deformities. Although this method was compared to the removable mandibular retractor in terms of skeletal and dentoalveolar changes, but the published paper did not report any information about the associated levels of pain and discomfort as well the general acceptability to this treatment modality.

ELIGIBILITY:
Inclusion Criteria:

1. Class III malocclusion according to Angle
2. Presence of anterior cross bite on two teeth or more
3. Class III Skeletal relationship confirmed radiographically (-4<ANB<+1)
4. The lower incisors have normal inclination (Incisor-Mandibular-Plane angle not exceeding 100° and not less than 85°)
5. Late mixed dentition or the beginning of the permanent dentition
6. Eruption of The lower canines and first premolars on both sides
7. Absence of craniofacial syndromes or cleft lip and/or palate abnormalities
8. no supernumerary teeth or missing teeth except for the third molars
9. no previous orthodontic treatment

Exclusion Criteria:

1. Pure maxillary deficiency
2. Pure mandibular prognathism
3. Diseases that prevent the application of mini-implants (e.g. Osteoporosis- cortisone and its derivatives treatment - radiation)
4. The roots of the canine are so close to the first premolar
5. Long face (Maxillary-mandibular plane angle greater than 30° or Mandibular-Cranial-Base angle greater than 36°).

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2015-02-15 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2016-05-10 (Actual)

PRIMARY OUTCOMES:
Change in the sensation of tension or pressure | Questionnaires will be filled at the following assessment times: one day following appliance insertion (T1), one week (T2), six weeks (T3), three months (T4) and after 6 months of appliance insertion (T5)
  Patients will be asked this question about their sensation of tension or pressure (Item no 01):
  Do you have a sense of tension and pressure in your soft tissues?
  A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the first six months of treatment.
  A four-point Likert scale is going to be used consisting of: (not at all), (little), (much) or (very much) to which points 0, 1, 2 and 3 respectively are going to be ascribed. Each questionnaire is going to be completed by the child in the presence of one of his/her parents.
Change in the perception of pain | Questionnaires will be filled at the following assessment times: one day following appliance insertion (T1), one week (T2), six weeks (T3), three months (T4) and after 6 months of appliance insertion (T5)
  Patients will be asked this question about their perception of pain (Item no 02):
  'Have you experienced any degree of pain?'
  A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the first six months of treatment. A four-point Likert scale is going to be used consisting of: (not at all), (little), (much) or (very much) to which points 0, 1, 2 and 3 respectively are going to be ascribed. Each questionnaire is going to be completed by the child in the presence of one of his/her parents.
Change in the perception of speech | Questionnaires will be filled at the following assessment times: one day following appliance insertion (T1), one week (T2), six weeks (T3), three months (T4) and after 6 months of appliance insertion (T5)
  Patients will be asked this question about any change encountered in the articulation of sounds (Item no 03):
  'Do you feel that your articulation has changed?'
  A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the first six months of treatment. A four-point Likert scale is going to be used consisting of: (not at all), (little), (much) or (very much) to which points 0, 1, 2 and 3 respectively are going to be ascribed. Each questionnaire is going to be completed by the child in the presence of one of his/her parents.
Change in swallowing ability | Questionnaires will be filled at the following assessment times: one day following appliance insertion (T1), one week (T2), six weeks (T3), three months (T4) and after 6 months of appliance insertion (T5)
  Patients will be asked this question about any difficulties encountered during swallowing (Item no 04):
  'Do you have difficulty in swallowing?'
  A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the first six months of treatment. A four-point Likert scale is going to be used consisting of: (not at all), (little), (much) or (very much) to which points 0, 1, 2 and 3 respectively are going to be ascribed. Each questionnaire is going to be completed by the child in the presence of one of his/her parents.
Change in mandibular restriction | Questionnaires will be filled at the following assessment times: one day following appliance insertion (T1), one week (T2), six weeks (T3), three months (T4) and after 6 months of appliance insertion (T5)
  Patients will be asked this question about any restrictions encountered in lower jaw movements (Item no 05):
  'Do you have a sense of your mandible movement being restricted?'
  A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the first six months of treatment. A four-point Likert scale is going to be used consisting of: (not at all), (little), (much) or (very much) to which points 0, 1, 2 and 3 respectively are going to be ascribed. Each questionnaire is going to be completed by the child in the presence of one of his/her parents.
Change in self-confidence perception | Questionnaires will be filled at the following assessment times: one day following appliance insertion (T1), one week (T2), six weeks (T3), three months (T4) and after 6 months of appliance insertion (T5)
  Patients will be asked this question about their feelings when meeting other people regarding self-confidence (Item no 06):
  'Do you have any feeling of embarrassment or lack of confidence?'
  A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the first six months of treatment. A four-point Likert scale is going to be used consisting of: (not at all), (little), (much) or (very much) to which points 0, 1, 2 and 3 respectively are going to be ascribed. Each questionnaire is going to be completed by the child in the presence of one of his/her parents.

CONTACTS AND LOCATIONS:
Overall Officials: Abdulmalek MR Majanni, DDS MSc, Principal Investigator — PhD student, Orthodontics Department, University of Damascus Dental School; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Associate Professor of Orthodontics, University of Damascus Dental School
Locations (1):
- Orthodontic Department, University of Hama Dental School, Hama, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sergl HG, Klages U, Zentner A. Pain and discomfort during orthodontic treatment: causative factors and effects on compliance. Am J Orthod Dentofacial Orthop. 1998 Dec;114(6):684-91. doi: 10.1016/s0889-5406(98)70201-x. PMID 9844209
- [Background] Khattab TZ, Farah H, Al-Sabbagh R, Hajeer MY, Haj-Hamed Y. Speech performance and oral impairments with lingual and labial orthodontic appliances in the first stage of fixed treatment. Angle Orthod. 2013 May;83(3):519-26. doi: 10.2319/073112-619.1. Epub 2012 Oct 18. PMID 23075062
- [Background] Idris G, Hajeer MY, Al-Jundi A. Acceptance and discomfort in growing patients during treatment with two functional appliances: a randomised controlled trial. Eur J Paediatr Dent. 2012 Sep;13(3):219-24. PMID 22971260
- [Background] Saleh M, Hajeer MY, Al-Jundi A. Assessment of pain and discomfort during early orthodontic treatment of skeletal Class III malocclusion using the Removable Mandibular Retractor Appliance. Eur J Paediatr Dent. 2013 Jun;14(2):119-24. PMID 23758461
- [Background] Gibreal O, Hajeer MY, Brad B. Evaluation of the levels of pain and discomfort of piezocision-assisted flapless corticotomy when treating severely crowded lower anterior teeth: a single-center, randomized controlled clinical trial. BMC Oral Health. 2019 Apr 16;19(1):57. doi: 10.1186/s12903-019-0758-9. PMID 30991984